CLINICAL TRIAL: NCT02508493
Title: Validation of the THINC-it Tool for Cognitive Dysfunction in Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Brain and Cognition Discovery Foundation (Other)
Collaborators: Co-Principal Investigators: Dr. Roger S. McIntyre & Dr. John Harrison (Unknown); Imperial College London (Other)
Responsible Party: Principal Investigator, Roger McIntyre, Executive Director, Brain and Cognition Discovery Foundation
Other Study IDs: BCDF-THINC.it
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major Depressive Disorder Population: 100 Individuals with DSM-5-defined MDD, aged 18-65
  Interventions: Other: THINC-it Tool; Other: Pencil-and-paper Cognitive Tests
- Healthy Control Population: 100 healthy controls matched on age, sex and years of education
  Interventions: Other: THINC-it Tool; Other: Pencil-and-paper Cognitive Tests

INTERVENTIONS:
Other: THINC-it Tool — Digitalized cognitive test application administering the following cognitive test components:
  * Digit Symbol Substitution Test (DSST)
  * Choice Reaction Time (CRT)
  * One-back working memory tool
  * Trail Making Test B (TMT-B)
  * Perceived Deficits Questionnaire-5 Depression (PDQ-5-D)
Other: Pencil-and-paper Cognitive Tests — Pencil-and-paper versions of the following cognitive tests:
  * Digit Symbol Substitution Test (DSST)
  * Trail Making Test B (TMT-B)
  * Perceived Deficits Questionnaire-5 Depression (PDQ-5-D)
  * Variant of Choice Reaction Time (CRT)
  * Variant of the One-back working memory tool

SUMMARY:
Cognitive dysfunction is a highly persistent, pervasive and progressive abnormality in young adults (i.e., 18-65 years) with MDD. It has also been shown that among adults with MDD who are gainfully employed, measures of cognition are a greater determinant of overall workplace performance than is total depression symptom severity. Several lines of evidence indicate that cognitive deficits that persist between episodes of depression are critical determinants of functional recovery in the workplace. The functional implications associated with cognitive impairment provide the impetus for systematic evaluation, measurement and assessment of the domains of cognition expected to be impaired in this patient population.

To date, no measurement tool has been sufficiently validated and/or determined to be sensitive to the cognitive deficits in younger adults with MDD. Major limitations of available comprehensive psychometric tools include relative lack of availability, cost, lack of access to most healthcare providers, and above all else, the lengthy time to administer. Moreover, the need for a psychometrist to interpret the results adds to the complexity and the costliness of such an endeavor.

It is imperative that any tool recommended for clinical utility be aligned with the busy nature of a high-volume clinical practice. The ideal gold standard tool for assessing the presence of cognitive dysfunction in MDD in the clinical environment should include, but not be limited to, features such as good conceptual coverage of cognitive domains affected in MDD, good sensitivity and reliability, and it should be relatively uninfluenced by culture effects and practice effects. The tool would also need to be brief, easy to administer and interpret, and complement busy clinical practice.

This study is designed to validate a brief user-friendly tool capable of detecting deficit in cognitive performance among adults with MDD. Data will be gathered with the aim to determine whether the proposed tool identifies cognitive deficits in adults with MDD and differentiates the clinical MDD population from healthy controls.

It is anticipated that the THINC-it tool will be free of charge and downloadable from the THINC-it website for use in the primary care and specialty setting. The THINC-it tool will be accessible via computers/tablets, will take 20 minutes to self-administer in a clinical setting, and the performance results will be immediately available.

ELIGIBILITY:
MDD Population:

Inclusion Criteria:

* That participant is able and willing to provide informed consent.
* The participant is male or female between the ages of 18-65.
* The participant has received a diagnosis of a major depressive disorder (MDE) as per DSM-5 criteria.
* Current MDE is confirmed by the MINI for DSM-IV-TR.
* The participant is an outpatient at a psychiatric setting.
* The participant has a MADRS score equal to or greater than 22.
* The reported duration of current depressive episode is at least 3 months.
* The participant has been receiving a stable antidepressant dose for a minimum of 2 weeks prior to the study visit.
* At least one prior episode by history of depression validated by previous treatment (e.g. guidelines-informed pharmacotherapy and/or manual-based psychotherapy).
* Health Canada-approved antidepressant; add-on agents commensurate with Canadian (i.e. CANMAT) and American treatment-guidelines for MDD will be permitted.
* Enrollment in manual-based and/or supportive psychotherapy will be permitted.

Exclusion Criteria:

* Current alcohol and/or substance use disorder.
* Presence of comorbid psychiatric disorder other than MDD that is a focus of clinical concern as confirmed by the MINI for DSM-IV-TR.
* Medications approved for and/or employed off label for cognitive dysfunction (e.g. psychostimulants).
* Any medication for a general medical disorder that in the opinion of the investigator may affect cognitive function (e.g. corticosteroids, beta-blockers).
* Use of benzodiazepines within 12 hours of THINC-it tool administration.
* Consumption of alcohol within 8 hours of THINC-it tool administration.
* The patient has physical, cognitive, or language impairment of some severity as to adversely affect the validity of the data derived from neuropsychological tests.
* The patient is diagnosed with a reading disability or dyslexia.
* The patient cannot have a clinically significant learning disorder by history.
* The patient has received electroconvulsive therapy (ECT) in the last 6 months.
* The patient has a history of moderate or severe head trauma (e.g. loss of consciousness for over 1 hour), other neurological disorders, or unstable systemic medical diseases that in the opinion of the investigator are likely to affect the central nervous system.

Healthy Controls:

Inclusion Criteria:

* No current or past history of mental disorder as evidence by MINI or DSM-IV-TR.
* No first-degree relative with an established diagnosis by a healthcare provider of a mood or psychiatric disorder.
* No unstable medical disorders.

Exclusion Criteria:

* Any medication for a general medical disorder that in the opinion of the investigator may affect cognitive function (e.g. corticosteroids, beta-blockers).
* Consumption of alcohol within 8 hours of THINC-it tool administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients will be enrolled at a single site, located in Toronto, Ontario, Canada. The total planned number of participants is:
  * 100 individuals with DSM-5-defined MDD, aged 18-65
  * 100 healthy controls matched on age, sex and years of education An equal allocation of subjects with MDD between the ages of 18-44 and 45-65 will be enrolled.
  Healthy controls will be consecutively recruited via media announcements.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composite THINC-it Tool Score | up to1 week
  The composite THINC-it tool score is the integrated total score of results from performance on five sub-component cognitive tests of the THINC-it tool.
Digit Symbol Substitution Test (DSST) - THINC-it tool version | Up to 1 week
Choice Reaction Time (CRT) - THINC-it tool version | Up to 1 week
One-back working memory test - THINC-it tool version | Up to 1 week
Trail Making Test B - THINC-it tool version | Up to 1 week
Perceived Deficits Questionnaire 5 item for depression (PDQ-5-D) - THINC-it tool version | Up to 1 week
Digit Symbol Substitution Test (DSST) - Pencil-and-paper version | Up to 1 week
Choice Reaction Time (CRT) - Pencil-and-paper version | Up to 1 week
One-back working memory test - Pencil-and-paper version | Up to 1 week
Trail Making Test B - Pencil-and-paper version | Up to 1 week
Perceived Deficits Questionnaire 5 item for depression (PDQ-5-D) - Pencil-and paper version | Up to 1 week

SECONDARY OUTCOMES:
Endicott Workplace Productivity Scale (EWPS) | Up to 1 week
Sheehan Disability Scale (SDS) | Up to 1 week
Pittsburgh Sleep Quality Index (PSQI) | Up to 1 week
Clinical Global Impression (CGI) | Administered at one timepoint to healthy controls and to subjects with MDD after administration of primary cognitive test instruments.
Montgomery Asberg Depression Rating Scale (MADRS) | Up to 1 week
Generalized Anxiety Disorder 7-Item (GAD-7) | Administered at one timepoint to healthy controls and to subjects with MDD after administration of primary cognitive test instruments.
WHO-5 Well-being Index (WHO-5) | Up to 1 week
Visual Analog Scale (VAS) | Up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, Principal Investigator — Brain and Cognition Discovery Foundation
Locations (1):
- CRTCE/KJK Healthplex, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cha DS, Carmona N, Cha RH, Zhou AJ, Subramaniapillai M, Mansur RB, Lee Y, Lee JH, Lee J, Almatham F, Alageel A, Rosenblat JD, Shekotikhina M, Rong C, Harrison J, McIntyre RS. Perceived sleep quality predicts cognitive function in adults with major depressive disorder independent of depression severity. Ann Clin Psychiatry. 2019 Feb;31(1):17-26. PMID 30372511
- [Derived] Cha DS, Carmona NE, Rodrigues NB, Mansur RB, Lee Y, Subramaniapillai M, Phan L, Cha RH, Pan Z, Lee JH, Lee J, Almatham F, Alageel A, Rosenblat JD, Shekotikhina M, Rong C, Harrison J, McIntyre RS. Cognitive impairment as measured by the THINC-integrated tool (THINC-it): The association with self-reported anxiety in Major Depressive Disorder. J Affect Disord. 2018 Oct 1;238:228-232. doi: 10.1016/j.jad.2018.05.006. Epub 2018 Jun 1. PMID 29886204
- [Derived] Carmona NE, Subramaniapillai M, Mansur RB, Cha DS, Lee Y, Fus D, McIntyre RS. Sex differences in the mediators of functional disability in Major Depressive Disorder. J Psychiatr Res. 2018 Jan;96:108-114. doi: 10.1016/j.jpsychires.2017.09.025. Epub 2017 Sep 30. PMID 28992527
- [Derived] McIntyre RS, Best MW, Bowie CR, Carmona NE, Cha DS, Lee Y, Subramaniapillai M, Mansur RB, Barry H, Baune BT, Culpepper L, Fossati P, Greer TL, Harmer C, Klag E, Lam RW, Wittchen HU, Harrison J. The THINC-Integrated Tool (THINC-it) Screening Assessment for Cognitive Dysfunction: Validation in Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jul;78(7):873-881. doi: 10.4088/JCP.16m11329. PMID 28858441